CLINICAL TRIAL: NCT06256692
Title: Hypoxemia in the First 24 Hours After Trauma - an Observational Study
Acronym: HYPOX24
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other); Laegeforeningens Forskningsfond (Unknown)
Responsible Party: Principal Investigator, Jacob Steinmetz, MD, professor, Rigshospitalet, Denmark
Other Study IDs: p-2023-15008; H-23065206 (Other: Research Ethics Committee, Capital Region, Denmark)
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Trauma; Trauma Injury; Hypoxemia; Hypoxia; Oxygen Deficiency
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pulse oximeter — No real intervention, but all study participants will have an additional pulse oximeter attached, to measure oxygen saturation.

SUMMARY:
The goal of this observational study is to investigate the occurrence of hypoxemia (an abnormally low concentration of oxygen in the blood) in trauma patients within the first 24 hours of hospital admission following arrival to a trauma center.

The main questions the study aims to answer are:

* Do trauma patients experience hypoxemia during the initial 24 hours of hospital admission following trauma?
* What is the daily distribution of potential hypoxemic episodes?

The investigators expect that hypoxemic episodes will be more frequent during the night (20.00-07.59) than during the day (08.00-19.59)

An additional pulse oximeter will be attached to the participants, which measures oxygen saturation in the blood during the first 24 hours of hospital admission after trauma.

DETAILED DESCRIPTION:
Trauma is one of the leading causes of death and disability on a global scale. Advanced Trauma Life Support guidelines state serious concern with the appearance of hypoxemia after trauma, and consequently recommend that supplemental oxygen should be provided for all severely injured trauma patients to avoid hypoxemia in the initial phase. Oxygen is a vital part of human physiology and must be delivered to all metabolically active cells in the body. When patients receive supplemental oxygen, a series of autoregulatory mechanisms happen to ensure optimal oxygen levels and prevent hypoxemia and hyperoxemia which can have different harmful effects. The lack of oxygen resulting in hypoxemia can potentially be a reversible cause of poor outcomes and in worst case death, hence supplemental oxygen is recommended for trauma patients, although the evidence is sparse.

In other high-risk patient groups, such as surgical and chronic obstructive pulmonary disease (COPD) patients, a study monitored arterial oxygen saturation (SpO2) continuously and found that cumulative duration of desaturations with SpO2 < 85% was significantly associated with myocardial injury after both surgery and exacerbation of COPD. In stroke patients, a study found a higher mortality in patients that experienced hypoxemia, but after adjusting for National Institute of Health Stroke Scale and age, this association was not significant. In the study, hypoxemia was found at all stages during admission. Using continuous monitoring for 48 hours a study found that hypoxemia was common and prolonged in patients recovering from noncardiac surgery. Furthermore, this study showed that 90% of hypoxemic episodes SpO2 < 90% for at least one hour went undetected by standard spot checks, which were typically conducted at intervals of 4-6 hours.

Trauma patients can also be characterized as high-risk patients due to a high mortality. The incidence of prehospital hypoxemia in traumatic brain injury patients has been studied, a study found a prevalence of 37.9%,11 and another study discovered that prehospital hypoxemia was associated with higher mortality. Evidence about the incidence of hypoxemia in trauma patients after admission to a hospital is not well established. There is reason to suspect that trauma patients can experience episodes of hypoxemia after admission and that the incidence of hypoxemia may differ between day and night as shown in several other patient populations. Potential incidences of severe hypoxemia, from patients being admitted to a trauma centre to subsequent care in a ward, should be avoided, since severe hypoxemia is associated with harmful effects. Hypoxemia can be detected and potentially corrected with more advanced measuring equipment. It is relevant to conduct a study with the purpose of determining the occurrence and distribution over the first 24 hours after hospital admission of hypoxemia by continuous SpO2 monitoring in trauma patients, since this could potentially have important clinical implications and be useful in improving patient outcomes.

This study is a single centre study of trauma patients at Rigshospitalet, Denmark. Rigshospitalet holds the only major trauma centre in the eastern part of Denmark, and every year around 1000 trauma patients are treated here. Patients are admitted from the Capital Region of Denmark with around 1.9 million inhabitants and the Region of Zealand with around 850.000 inhabitants.

All patients with trauma team activation in the trauma bay at Rigshospitalet, including both direct transport and secondary transfers, will be screened for potential inclusion in the study.

The trauma bay at Rigshospitalet will be equipped with the oximetry equipment, and measurement can be started as early as possible. At the trauma bay, a doctor will conduct the screening and inclusion of patients to the study at arrival. After study inclusion, monitoring equipment will be attached by a nurse in the trauma bay. Subsequently a member of the study investigator group will obtain consent.

Continuous pulse oximetry will be used to measure SpO2. SpO2, heart rate, pulse amplitude and alarm status will be measured every second during a 24-hour period on all study participants.

The Nellcor™ Portable SpO2 Patient Monitoring System, PM10N (Medtronic, 15 Hampshire Street, Mansfield, MA 02048, USA) is used as monitoring device. The Covidien Nellcor FLEXMAX or a similar probe will be placed on the patients' index finger, alternatively another finger or toe.

Data collection will continue for up to 24 hours. If there is an untimely removal of the probe, the device will switch of, and data collection will stop at this point, unless the device is turned on again. After 24 hours of measurement, an investigator will collect the device and transfer the data by USB cable to a computer for secure storage and further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Blunt or penetrating mechanism of trauma
* Trauma team activation
* Admission to a ward/ICU from trauma centre

Exclusion Criteria:

* Patients with a suspicion of carbon monoxide intoxication
* No applicable finger or toe for sensor attachment
* Trauma team activation was cancelled
* No available pulse oximeter at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with trauma team activation in the trauma bay at Rigshospitalet, including both direct transport and secondary transfers, will be screened for potential inclusion in the study. Patients will be included if they comply with the above eligibility criteria
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of hypoxemia | 24 hours
  The occurrence and daily distribution of clinically relevant hypoxemic episodes defined as SpO2 <90% for >5 minutes, within the first 24 hours after trauma

SECONDARY OUTCOMES:
Location of hypoxemia (Specific departments) | 24 hours
  The location of the occurrence of clinically relevant hypoxemic episodes SpO2 < 90% > 5 minutes in specific departments including trauma centre, ICU, general ward, operating theatre and recovery room.
Prolonged hypoxemic episodes | 24 hours
  The occurrence of prolonged hypoxemic episodes SpO2 < 90% for > 30 minutes per episode
Cumulated time of hypoxemia | 24 hours
  Cumulated time of hypoxemia SpO2 <90%

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Steinmetz, MD,professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Region H, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zulazmi NA, Arulsamy A, Ali I, Zainal Abidin SA, Othman I, Shaikh MF. The utilization of small non-mammals in traumatic brain injury research: A systematic review. CNS Neurosci Ther. 2021 Apr;27(4):381-402. doi: 10.1111/cns.13590. Epub 2021 Feb 4. PMID 33539662
- [Background] ATLS Subcommittee; American College of Surgeons' Committee on Trauma; International ATLS working group. Advanced trauma life support (ATLS(R)): the ninth edition. J Trauma Acute Care Surg. 2013 May;74(5):1363-6. doi: 10.1097/TA.0b013e31828b82f5. No abstract available. PMID 23609291
- [Background] Rhodes CE, Denault D, Varacallo MA. Physiology, Oxygen Transport. 2022 Nov 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538336/ PMID 30855920
- [Background] Lopez-Barneo J, Ortega-Saenz P, Gonzalez-Rodriguez P, Fernandez-Aguera MC, Macias D, Pardal R, Gao L. Oxygen-sensing by arterial chemoreceptors: Mechanisms and medical translation. Mol Aspects Med. 2016 Feb-Mar;47-48:90-108. doi: 10.1016/j.mam.2015.12.002. Epub 2015 Dec 18. PMID 26709054
- [Background] Singer M, Young PJ, Laffey JG, Asfar P, Taccone FS, Skrifvars MB, Meyhoff CS, Radermacher P. Dangers of hyperoxia. Crit Care. 2021 Dec 19;25(1):440. doi: 10.1186/s13054-021-03815-y. PMID 34924022
- [Background] Eskesen TG, Baekgaard JS, Steinmetz J, Rasmussen LS. Initial use of supplementary oxygen for trauma patients: a systematic review. BMJ Open. 2018 Jul 6;8(7):e020880. doi: 10.1136/bmjopen-2017-020880. PMID 29982208
- [Background] Loft FC, Rasmussen SM, Elvekjaer M, Haahr-Raunkjaer C, Sorensen HBD, Aasvang EK, Meyhoff CS; WARD-Project Group. Continuously monitored vital signs for detection of myocardial injury in high-risk patients - An observational study. Acta Anaesthesiol Scand. 2022 Jul;66(6):674-683. doi: 10.1111/aas.14056. Epub 2022 Mar 14. PMID 35247272
- [Background] Rowat AM, Dennis MS, Wardlaw JM. Hypoxaemia in acute stroke is frequent and worsens outcome. Cerebrovasc Dis. 2006;21(3):166-72. doi: 10.1159/000090528. Epub 2005 Dec 23. PMID 16388191
- [Background] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Background] Murdock D. Trauma: when there's no time to count. AORN J. 2008 Feb;87(2):322-8. doi: 10.1016/j.aorn.2007.07.008. PMID 18323023
- [Background] Stassen W, Welzel T. The prevalence of hypotension and hypoxaemia in blunt traumatic brain injury in the prehospital setting of Johannesburg, South Africa: A retrospective chart review. S Afr Med J. 2014 May 12;104(6):424-7. doi: 10.7196/samj.7494. PMID 25214252
- [Background] Chi JH, Knudson MM, Vassar MJ, McCarthy MC, Shapiro MB, Mallet S, Holcroft JJ, Moncrief H, Noble J, Wisner D, Kaups KL, Bennick LD, Manley GT. Prehospital hypoxia affects outcome in patients with traumatic brain injury: a prospective multicenter study. J Trauma. 2006 Nov;61(5):1134-41. doi: 10.1097/01.ta.0000196644.64653.d8. PMID 17099519
- [Background] Ali K, Cheek E, Sills S, Crome P, Roffe C. Day-night differences in oxygen saturation and the frequency of desaturations in the first 24 hours in patients with acute stroke. J Stroke Cerebrovasc Dis. 2007 Nov-Dec;16(6):239-44. doi: 10.1016/j.jstrokecerebrovasdis.2007.07.004. PMID 18035240
- [Background] Fanfulla F, Grassi M, Taurino AE, D'Artavilla Lupo N, Trentin R. The relationship of daytime hypoxemia and nocturnal hypoxia in obstructive sleep apnea syndrome. Sleep. 2008 Feb;31(2):249-55. doi: 10.1093/sleep/31.2.249. PMID 18274273
- [Background] Galatius-Jensen S, Hansen J, Rasmussen V, Bildsoe J, Therboe M, Rosenberg J. Nocturnal hypoxaemia after myocardial infarction: association with nocturnal myocardial ischaemia and arrhythmias. Br Heart J. 1994 Jul;72(1):23-30. doi: 10.1136/hrt.72.1.23. PMID 8068464
- See also: Data from Traumacentre — http://www.rigshospitalet.dk/afdelinger-og-klinikker/hovedorto/traumecenter-og-akut-modtagelse/om-traumecentret/Sider/tal-og-fakta.aspx
- See also: Link on statistics — http://www.statbank.dk/FOLK1A